CLINICAL TRIAL: NCT05474170
Title: Impact of 2 Resuscitation Sequences on Alveolar Ventilation During the First Minute of Simulated Pediatric Cardiac Arrest: Randomized Cross-Over Trial
Brief Title: Impact of 2 Resuscitation Sequences on Management of Simulated Pediatric Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneve TEAM Ambulances (Other)
Collaborators: Service de la protection et de la sécurité, Neuchâtel (Unknown); École supérieure de soins ambulanciers, Genève (Unknown); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stuby Loric, Principal Investigator, Geneve TEAM Ambulances
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPR-AHA/ERC
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiopulmonary Arrest; Pediatric ALL; Resuscitation
MeSH Terms: conditions — Heart Arrest; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data extraction will be fully automated and the statistician will not know the identity of the participants or the sequence they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AHA --> ERC (Experimental): This group will first apply the AHA resuscitation sequence, then the ERC one
  Interventions: Other: AHA resuscitation sequence; Other: ERC resuscitation sequence
- ERC --> AHA (Active Comparator): This group will first apply the ERC resuscitation sequence, then the AHA one
  Interventions: Other: AHA resuscitation sequence; Other: ERC resuscitation sequence

INTERVENTIONS:
Other: AHA resuscitation sequence — Starting the cardiopulmonary resuscitation by following the AHA guideline, meaning starting with 15 chest compressions, followed by 2 ventilations
Other: ERC resuscitation sequence — Starting the cardiopulmonary resuscitation by following the ERC guideline, meaning starting with 5 initial ventilations, then alternating 15 chest compressions with 2 ventilations

SUMMARY:
The International Liaison Committee on Resuscitation regularly publishes a Consensus on Science with Treatment Recommendations but guidelines can nevertheless differ when knowledge gaps persist. In case of pediatric cardiac arrest, the American Heart Association recommends following the adult resuscitation sequence i.e., starting with chest compressions. Conversely, the European Resuscitation Council advocates the delivery of 5 initial rescue breaths before starting chest compressions. Carrying out a randomized trial in children in cardiac arrest to assess the impact of these strategies would prove particularly challenging and ethical concerns may prevent such a trial from being performed. This will be a superiority, cross-over randomized trial whose goal is to determine the impact of these 2 resuscitation sequences on alveolar ventilation in a pediatric model of cardiac arrest. While not definitive, its results could help fill part of the current knowledge gap.

DETAILED DESCRIPTION:
This will be a randomized, cross-over, superiority trial. The intention is to carry it out on the first Prehospital Research Day which will be held on September 1st, 2022, i.e., on a single date. This event will take place at a single center in Neuchâtel, Switzerland. If the intended sample size cannot be reached on this day, or if technical issues prevent data from being collected or extracted, other study sites will be considered.

Participant recruitment will be conducted online. A web-based platform based on the Joomla 4 (Open Source Matters, New York, USA) content management system will be specifically created for the purpose of this study. The Event Booking 4 component (Joomdonation, Hanoi, Vietnam) will be used to create 20-minute time slots. Demographic data will be collected during the registration process. Consent will be gathered electronically.

Since the objective of this study is to assess the impact of basic airway management and ventilation maneuvers only, there will be no stratification since all the professionals eligible for inclusion should be equally proficient in basic airway management. Furthermore, all participants will be able to practice this skill on a manikin identical to the one used to perform the study. This training will not be time limited and will take place immediately before the sequence during which data will be collected.

An investigator who will not be present during the resuscitation sequences will create stacks of opaque, sealed envelopes. Each stack of 10 envelopes will contain an equal number of American Heart Association (AHA) and European Resuscitation Council (ERC) allocations. Randomization will take place after the training session. The first leader will choose and open one of the envelopes placed on a table in random order by one of the on-site investigators. This will determine the resuscitation sequence which will first be used by the team.

A SimBaby manikin (Laerdal SimBaby, Laerdal Medical, Stavanger, Norway) will be used in this study. The SimBaby is a realistic manikin representing a 9-month-old infant. The manikin weighs 4.9 kg and is 71 cm tall. It is accompanied with a dedicated multiparameter monitor/defibrillator. Back compensation, using a folded blanket, will be applied. An appropriately sized bag-valve-mask (BVM) device will be ready for use next to the manikin. The defibrillation pads will be already attached.

Participants will be told that they are facing a 9-month old infant who suddenly collapsed. They will be told that there is no foreign body airway obstruction and that the infant is in cardiac arrest.

Each team of two people will perform 4 resuscitation sequences of one minute each. Each participant will act as leader for two successive resuscitation sequences, the first of which will be carried out according to the random allocation described above. The scenario will be identical for all resuscitation sequences. After completing these two sequences, participants will exchange their roles, and the new leader will pick up another opaque, sealed envelope. The content of this envelope will determine the resuscitation sequence the newly appointed leader will have to use first.

The timer will start (T0) at the moment when the first action (chest compression or ventilation) will have been performed and will stop exactly after 60 seconds.

It will not be possible to blind the participants or the on-site investigators as to the design of the study or even to the allocation of the participants. Nevertheless, the outcomes will not be communicated to the participant. In addition, data extraction will be fully automated and the statistician will not know the identity of the participants or the sequence they were allocated to.

ELIGIBILITY:
Inclusion Criteria:

* Being issued from one of the following profession: Emergency medical technicians (EMTs), paramedics, nurses and physicians

Exclusion Criteria:

* Being member of the study team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Alveolar ventilation | 1 minute
  The alveolar ventilation will be determined by subtracting the dead space volume from each ventilation. According to the appropriate Best Guess formula, a 9-month old infant should weigh around 9 kg (0.5 x age in months + 4.5). Using the formula proposed by Numa and Newth, this corresponds to a dead space of around 25 ml.

SECONDARY OUTCOMES:
The total number of ventilations | 1 minute
  This will be the count of the number of ventilations delivered during the scenario
The proportion of ventilations within, above and below the target volume | 1 minute
  According to the manikin's manufacturer, the target is 30 to 70 ml
The alveolar ventilation obtained without taking ventilation volumes over 70 ml into account | 1 minute
  This is similar to the primary outcome, but for this analysis, all ventilations will be individually capped at 45 ml
The proportion of compressions of correct depth | 1 minute
  The chest compression will be considered correct if ≥ 4.3 cm, corresponding to one third of the height of the manikin's chest i.e., 13 cm)
The proportion of chest compressions within, above and below the target rate. | 1 minute
  According to the guidelines, the target is 100 to 120 compressions per minute
The chest compression fraction (CCF) | 1 minute
  This corresponds to the time with compressions on the total time of the cardiopulmonary resuscitation sequence
The proportion of compressions with adequate chest recoil | 1 minute
  This corresponds to the proportion of compressions enough relaxed to let complete heart relaxation

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Suppan, MD, Principal Investigator — University of Geneva Hospitals and Faculty of Medicine
Locations (1):
- Swiss Prehospital Research Day, Neuchâtel, Canton of Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data set will be made publicly available on the Digital Commons Data repository
Time Frame: Data will be available after publication of the results
Access Criteria: Publicly available

REFERENCES:
- [Background] Suppan L, Jampen L, Siebert JN, Zund S, Stuby L, Ozainne F. Impact of Two Resuscitation Sequences on Alveolar Ventilation during the First Minute of Simulated Pediatric Cardiac Arrest: Randomized Cross-Over Trial. Healthcare (Basel). 2022 Dec 5;10(12):2451. doi: 10.3390/healthcare10122451. PMID 36553975
- See also: Whole project website — https://swiss-cpr-studies.ch/